CLINICAL TRIAL: NCT02700503
Title: Finding the Patient's Voice: Development of Practical Approaches for Adolescent and Family Focused Diabetes Prevention Programs
Brief Title: Finding the Patient's Voice Diabetes Prevention Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Indiana University Health (Other)
Responsible Party: Principal Investigator, Tamara S. Hannon, Associate Professor of Pediatrics, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1510313617
Record Dates: First submitted 2016-02-23; First posted 2016-03-07 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus, Type 2; Prediabetic State
Keywords: Diabetes prevention; type 2 diabetes; prediabetes; family
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Participants will be enrolled in the ENCOURAGE 2.0 family-based diabetes prevention intervention that was designed through our work in Aims 1 and 2 of the study. It is this modified population-level ENCOURAGE 2.0 family-based diabetes prevention intervention that will be studied.
  Interventions: Behavioral: Encourage 2.0

INTERVENTIONS:
Behavioral: Encourage 2.0 — Participants will be enrolled in the ENCOURAGE 2.0 family-based diabetes prevention intervention that was designed through our work in Aims 1 and 2 of the study. It is this modified population-level ENCOURAGE 2.0 family-based diabetes prevention intervention that will be studied.

SUMMARY:
This study uses patient engagement to develop a diabetes prevention program focused on adolescents and families.

DETAILED DESCRIPTION:
Due to increases in obesity, the onset of type 2 diabetes is occurring at an ever-younger age, and is associated with poor outcomes and rising costs, which emphasizes the need for prevention at earlier ages. To address this need, the investigators designed the ENCOURAGE Healthy Families curriculum; a program based on the scientifically proven U.S. Diabetes Prevention Program, and while data demonstrate a reduction in obesity and diabetes risk for mothers and their children, the investigators have encountered several barriers to widespread implementation, including:

1. helping youth/families understand the importance of prevention,
2. on-going interest and participation, and
3. differing personal beliefs.

Patient-centered research is needed to better understand what adolescents/families want in prevention initiatives, who should deliver program content, where and when to deliver programs in the community, and how adolescents/families wish to be informed of results. The investigators believe that by engaging patients and the community in the development process, the investigators will be able to obtain workable answers to these questions at a population level for high-risk youth/families in "real world" settings.

ELIGIBILITY:
Inclusion Criteria:

1. Overweight (BMI >85th percentile for age and sex, weight for height >85th percentile, or weight >120% of ideal [50th percentile] for height)
2. At least two of the following risk factors:

   * Have been diagnosed with prediabetes;
   * Have a family history of T2DM in first- and second-degree relatives;
   * Belong to a minority race/ethnic group (Native Americans, African-Americans, Hispanic Americans, Asians/South Pacific Islanders);
   * Have conditions associated with insulin resistance; and/or
   * Have had gestational diabetes or were exposed to gestational diabetes in utero.
3. A family support person who is also willing to participate in the study. This person would preferably be a parent also at risk for diabetes (history of gestational diabetes, prediabetes, or with T2D).

Exclusion Criteria:

1. Type 2 diagnosis

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 146 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Subject's BMI calculation Charted on CDC Stature for Age and Weight for Age Percentiles chart | 12 months

SECONDARY OUTCOMES:
Hemoglobin A1C | 12 months
Physical activity | 12 months
  self-report
Quality of life | 12 months
  Pediatric Quality of Life Inventory
Intervention group session attendance | 12 months
Dietary records | 12 months
  Semi-quantitative food frequency questionniare

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Hannon, MD, Principal Investigator — Indiana University
Locations (3):
- United States (3):
  - Riley Children's Specialties, Carmel, Indiana
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Riley Children's Hospital, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: Undecided
undecided